CLINICAL TRIAL: NCT01766063
Title: BETASLEEP - SLEEP Quality and Functional Health Status, Fatigue, Comorbidities and Therapeutic Algorithms Among BETAferon® Treated MS Patients
Brief Title: Investigating the Relationship Between Sleep, Quality of Life,Other Disorders and Therapies in MS Patients on Betaferon
Acronym: BetaSleep
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16352; BF1212DE (Other: Company internal)
Record Dates: First submitted 2012-12-07; First posted 2013-01-11 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Sleep; Quality of life; Observational study
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Interferon beta-1b (Betaferon, BAY 86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaferon, BAY 86-5046) — Patients will be followed-up for 24 months

SUMMARY:
The study aims to investigate the relationship between sleep quality, quality of life,other disorders and therapies in Multiple Sclerosis (MS) patients treated with Betaferon.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age with relapsing remitting multiple sclerosis or a clinically isolated syndrome and an expanded disability status scale score ≤5.
* Patients must be on treatment with Betaferon and tolerate Betaferon according to the investigator's evaluation, but should not have received Betaferon longer than six months.
* Written informed consent must be obtained

Exclusion Criteria:

* Patients who do not tolerate Betaferon according to the investigator's evaluation or have been treated with Betaferon for more than six months.
* Patients receiving any other disease modifying drug or MS specific treatments
* Contraindications of Betaferon described in the Summary of Product Characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with relapsing remitting multiple sclerosis (RRMS) or patients with a clinically isolated syndrome (CIS) with an Expanded Disability Status Scale (EDSS) score ≤5 who tolerate Betaferon according to the investigator's evaluation, but have not received Betaferon longer than six months. Participants will be recruited from private neurological offices and neurology departments throughout Germany.
  In this non-interventional observational study, the decision on the duration and dosage of treatment is solely at the discretion of the attending physician.
  The medication is prescribed at regular visits to the investigator's office. Commercially available product will be used to treat the patients.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-03-14 (Actual)

PRIMARY OUTCOMES:
Sleep quality will be assessed by the Pittsburgh Sleep Quality Index (PSQI) | up to 3 years
Fatique assessed by the Modified Fatigue Impact Scale (MFIS) | up to 3 years
Functional health status assessed by Short Form-36 (SF-36) | up to 3 years

SECONDARY OUTCOMES:
Daytime sleepiness is measured with the Epworth Sleepiness Scale (ESS) | up to 3 years
Depression and anxiety is measured with the Hospital anxiety and depression scale (HADS) | up to 3 years
Pain is measured with the Hamburg Pain Adjective List (Hamburger Schmerz Adjektiv Liste (HSAL) | up to 3 years
Severity of restless legs syndrome measured with the International Restless Legs Syndrome Study (IRLSS) group rating scale. | up to 3 years

OTHER OUTCOMES:
Safety variables will be summarized using descriptive statistics based on adverse events collection | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Germany

REFERENCES:
- [Derived] Kotterba S, Neusser T, Norenberg C, Bussfeld P, Glaser T, Dorner M, Schurks M. Sleep quality, daytime sleepiness, fatigue, and quality of life in patients with multiple sclerosis treated with interferon beta-1b: results from a prospective observational cohort study. BMC Neurol. 2018 Aug 24;18(1):123. doi: 10.1186/s12883-018-1113-5. PMID 30143019